CLINICAL TRIAL: NCT02413905
Title: Characterizing the Gut Microbiota Alteration Associated With Severe Acute Malnutrition
Status: Completed | Type: Observational
Sponsor: Institut Hospitalo-Universitaire Méditerranée Infection (Other)
Responsible Party: Sponsor
Other Study IDs: SAMGUT
Record Dates: First submitted 2015-03-30; First posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Severe Malnutrition; Malnutrition; Infant Nutrition Disorders; Child Nutrition Disorders; Kwashiorkor; Marasmus
MeSH Terms: conditions — Malnutrition; Infant Nutrition Disorders; Child Nutrition Disorders; Kwashiorkor; Protein-Energy Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Senegal: Stool samples on Children with and without severe acute malnutrition in Senegal recruited in 3 locations (Dakar, Dielmo and Ndiop)
  Interventions: Biological: Stool samples
- Niger: Stool samples Children with and without severe acute malnutrition in Niger recruited in Niamey
  Interventions: Biological: Stool samples

INTERVENTIONS:
Biological: Stool samples — Stool samples

SUMMARY:
The investigators performed two case-control studies in Niger and Senegal analysing fecal microbiota to characterize the specificity of the gut microbiota alteration associated with severe acute malnutrition (SAM).

DETAILED DESCRIPTION:
Fecal samples of cases (severe acute malnutrition (SAM) ascertained according to the WHO definition) and controls (asymptomatic healthy children ascertained by clinical and anthropometric criteria) were analysed by v3v4 16S rRNA sequencing, redox and pH measurement and using specific polymerase chain reaction targeting Methanobrevibacter smithii and Bacteroides thetaiotaomicron. Based on the literature and oxydative stress reported in SAM, the investigators tested if the proportion of aerotolerant prokaryotes is increased among gut prokaryotes enriched in SAM in comparison to prokaryotes enriched in controls. The investigators further linked this to fecal redox potential and assessed the total number of bacteria in feces by flux cytometry.

ELIGIBILITY:
Inclusion criteria:

* Children aged 0-59 months of varying nutritional status from Niamey (Niger) and Dakar (Senegal).

Exclusion Criteria:

* Absence of parent or patient consent, antibiotic administration <2 months before stool collection and insufficient fecal amount. Exclusion criteria for controls included any form of malnutrition, presence of fever, acute respiratory infection (cough), acute or chronic diarrhea in the previous 4 weeks. Symptoms and complications of malnutrition (cough, fever, diarrhoea, vomiting) nor other form of malnutrition (moderate to severe stunting and underweight) were not a reason of exclusion for cases since they are considered as direct consequence and part of severe acute malnutrition.

Max Age: 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from Niamey and Dakar, Senegal
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Aerotolerant Odds ratio (AOR) | 1 day (Participants were not followed as this is a case-contol study only clinical and anthropometric data and fecal samples were collected the day of inclusion)
  AOR = (number of aerotolerant prokaryotes enriched in the gut of children with SAM * number of obligate anaerobic prokaryotes enriched in controls)/(number of aerotolerant prokaryotes enriched in controls * number of obligate anaerobic prokaryotes enriched in children with SAM)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Million, Study Chair — Assistance publique des Hôpitaux de Marseille
Locations (2):
- Hopital National, Niamey, Niger
- Clinic Notre Dame de L'Esperance, Thiaroye, Dakar, Senegal